CLINICAL TRIAL: NCT06055608
Title: Advancing Transplantation Outcomes in Children (CTOT-41)
Brief Title: Advancing Transplantation Outcomes in Children
Acronym: ADVANTage
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT CTOT-41
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Kidney Transplant
Keywords: kidney transplant; belatacept; sirolimus
MeSH Terms: interventions — Sirolimus; Abatacept; Mycophenolic Acid; Tacrolimus; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- (Group 1): Belatacept+Sirolimus group (Experimental): Participants in this group will receive antithymocyte globulin (ATG) + steroid taper + belatacept + (tacrolimus bridge, day 0-14) with conversion to sirolimus (day 30 +/-14 days)
  Interventions: Drug: Sirolimus; Biological: Belatacept; Drug: Tacrolimus (Group1); Drug: Anti-Thymocyte Globulin (ATG)
- (Group 2): Tacrolimus + Mycophenolate Mofetil (MMF) group (Active Comparator): Participants in this group will receive anti-thymocyte globulin (ATG) + steroid taper + tacrolimus + MMF
  Interventions: Drug: Mycophenolate Mofetil; Drug: Anti-Thymocyte Globulin (ATG); Drug: Tacrolimus (Group 2)

INTERVENTIONS:
Drug: Sirolimus — Participants in Group 1 will transition to sirolimus therapy on day 14 (+/- 5 days) - weight <40 kg will receive 3mg/m^ 2, with maintenance dose of 1 mg/m^2 divided BID - weight >= 40kg will receive 6mg/m^ 2, with maintenance dose of 2 mg daily
  Other Names: AY 22-989; Rapamune; Rapamycin
  Arms: (Group 1): Belatacept+Sirolimus group
Biological: Belatacept — Belatacept will be administered as an intravenous infusion over 30 minutes. The belatacept dose for the study is 10 mg/kg on post-operative day (POD) 1, 5, 14, 28, 56, 84 for the first 3 months, followed by 5 mg/kg every 4 weeks (+/-4 days), starting on month 4 until month 24
  Other Names: Nulojix
  Arms: (Group 1): Belatacept+Sirolimus group
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil-MMF will be initiated at 600 mg/m^2 BID until tacrolimus is at therapeutic levels, then 450 mg/m^2 BID
  Other Names: CellCept; MMF
  Arms: (Group 2): Tacrolimus + Mycophenolate Mofetil (MMF) group
Drug: Tacrolimus (Group1) — Participants will receive Prograf® (tacrolimus), or generic, initiated at 0.1 mg/kg BID within 48 hours of transplantation to attain target trough levels. Participants in Group 1 will be transitioned to sirolimus 2-4 weeks post-transplant
  Other Names: FK-506; FR-900506; Prograf
  Arms: (Group 1): Belatacept+Sirolimus group
Drug: Anti-Thymocyte Globulin (ATG) — Participants will receive induction therapy with anti-thymocyte globulin (1.5 mg/kg/dose, maximum 125 mg) starting intraoperatively on day 0 and continuing on days 2 and 3 (total dose 4.5 mg/kg). Total dose may be extended to 6 mg/kg over 1-2 days for delayed graft function
Drug: Tacrolimus (Group 2) — Participants will receive Prograf® (tacrolimus), or generic, initiated at 0.1 mg/kg BID within 48 hours of transplantation to attain target trough levels
  Other Names: FK-506; FR-900506; Prograf
  Arms: (Group 2): Tacrolimus + Mycophenolate Mofetil (MMF) group

SUMMARY:
This is a pediatric kidney transplant study comparing the safety and efficacy of an immunosuppressive regimen of belatacept and sirolimus to tacrolimus and Mycophenolate Mofetil (MMF). Two hundred participants will be randomized (1:1) to one of two groups within 24 hours following the transplant procedure. The duration of the study from time of transplant to the primary endpoint is 12-24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Participant and/or parent/guardian must be able to understand and provide informed consent
2. Male or female, 13-20 years of age at time of enrollment
3. Candidate for primary renal allograft from a living or deceased donor
4. EBV IgG seropositive, defined as evidence of acquired immunity shown by the presence of IgG antibodies to viral capsid antigen (VCA) and EBV nuclear antigen (EBNA)
5. EBV VCA IgM seronegative OR EBV VCA IgM seropositive on two occasions at least 3 months apart and an undetectable EBV PCR result within 1 month prior to enrollment
6. If a female participant of childbearing potential, a negative pregnancy test prior to conducting any study procedures
7. If participant has reproductive potential, agrees to use Food and Drug Administration (FDA) approved methods of birth control for the duration of the study
8. Negative test result for latent tuberculosis infection by tuberculosis skin test (purified protein derivative [PPD]) or Tuberculosis (TB) blood test (interferon gamma release assay [IGRA] i.e., QuantiFERON, T- SPOT.TB) within 12 months
9. In the absence of contraindication, vaccinations must be up to date per the Centers for Disease Control and Prevention (CDC) Guidelines and Division of Allergy, Immunology, and Transplantation (DAIT) Guidance for Patients in Transplant Trials

Enrollment criteria for donor source and age will be expanded using a stepwise approach determined by safety monitoring. Expansion criteria will include recipients down to age 6 and living donors. Safety data from each step will be reviewed by the study team, DSMB and FDA. If no safety concerns are identified, inclusion criteria will be expanded.

Exclusion Criteria:

1. Inability or unwillingness to comply with study protocol
2. Active infection requiring treatment, or viremia
3. History of malignancy
4. Receipt of any licensed or investigational live attenuated vaccine(s) within 4 weeks of enrollment
5. Prior history of organ transplantation
6. Listed for multi-organ transplant (e.g. heart- kidney, liver-kidney, multivisceral- kidney, lung- kidney)
7. Active systemic autoimmune disease at time of enrollment
8. Idiopathic Focal Segmental Glomerulosclerosis (FSGS), Membranoproliferative Glomerulonephritis (MPGN), C3 glomerulopathy, or atypical Hemolytic Uremic Syndrome (HUS) suspected at risk for recurrence
9. Use of immunosuppressants, biologics (including IVIG), chronic corticosteroids or investigational drug(s) within 8 weeks of enrollment
10. Known bleeding disorder
11. Sustained platelet count < 75,000 cells/microliters within 3 months of enrollment
12. History of inherited hypercoagulability requiring therapy more than aspirin
13. Panel Reactive Antibody (cPRA) greater than 80 percent
14. Clinically significant unrepaired congenital heart disease causing hemodynamic compromise
15. Uncontrolled diagnosed psychiatric disorder or self-reported drug or alcohol abuse that, in the opinion of the investigator, would interfere with the participant's ability to comply with study requirements
16. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study

Randomization Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for randomization.

1. If EBV serology to meet enrollment criteria was performed within 8 weeks of receiving IVIG, EBV VCA IgG and EBV EBNA IgG seropositivity, confirmed between enrollment and time of transplant

Randomization Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for randomization.

1. Sustained WBC <1500 or >20,000 per microliter within 3 months of randomization
2. Sustained liver function tests (AST and/or ALT) > 2x normal within 3 months of randomization
3. Active systemic autoimmune disease at time of transplant
4. Known bleeding disorder
5. Sustained platelet count < 75,000 cells/microliters within 3 months of enrollment
6. Current (within 45 days) or historical anti-HLA antibody to the donor prior to randomization
7. Recent recipient of any licensed or investigational live attenuated vaccine(s) within 4 weeks of randomization
8. Panel Reactive Antibody (cPRA) greater than 80 percent at any point in time
9. If a female participant of childbearing potential, a positive pregnancy test within 48 hours of randomization (all female participants of childbearing potential must complete a pregnancy test within 48 hours of randomization)
10. Treatment with immunosuppressants within 8 weeks of randomization, except in the case of planned transplant standard of care
11. Treatment with biologics (including IVIG) within 8 weeks of randomization

Ages: 13 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-05-22 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of de novo Donor Specific Antibody (dnDSA) (central lab) OR decline in estimated glomerular filtration rate (eGFR) >7.5 mL/min/1.73m^2 (central lab) | At 96 weeks post-transplant

SECONDARY OUTCOMES:
Incidence of clinical biopsy proven allograft rejection (central lab) | Within 96 weeks post-transplant
Time to development of clinical biopsy proven allograft rejection (central lab) | Within 96 weeks post-transplant
Incidence of subclinical biopsy proven allograft rejection (central lab) | Within 96 weeks post-transplant
Time to development of subclinical biopsy proven allograft rejection (central lab) | Within 96 weeks post-transplant
Incidence of Post-Transplant Lymphoproliferative Disease (PTLD) | Within 96 weeks post-transplant
Time to development of the PTLD | Within 96 weeks post-transplant
Incidence of Grade 3 and above opportunistic infections bacterial, viral, fungal, pneumocystis pneumonia, or parasitic infections assessed as a composite | Within 96 weeks post-transplant
Time to development of Grade 3 and above opportunistic infections bacterial, viral, fungal, pneumocystis pneumonia, or parasitic infections assessed as a composite | Within 96 weeks post-transplant

CONTACTS AND LOCATIONS:
Overall Officials: David Briscoe, MD, Study Chair — Boston Children's Hospital: Pediatric Transplantation; Eileen Chambers, MD, Study Chair — Duke University Medical Center: Department of Pediatrics
Locations (20):
- United States (20):
  - University of Alabama at Birmingham (Site # 71038), Birmingham, Alabama
  - Children's Hospital of Los Angeles (Site #: 71036), Los Angeles, California
  - Cedars-Sinai Medical Center (Site #: 71026), Los Angeles, California
  - Mattel Children's Hospital, UCLA (Site #: 71012), Los Angeles, California
  - UCSD Rady Children's Hospital (Site #: 71037), San Diego, California
  - Children's Hospital of Colorado (Site #: 71019), Aurora, Colorado
  - Nemours Children's Health (Site #: 71042), Wilmington, Delaware
  - Children's National Medical Center (Site #: 71039), Washington D.C., District of Columbia
  - Ann and Robert H. Lurie Children's Hospital of Chicago (Site #: 71016), Chicago, Illinois
  - Johns Hopkins Children's Center (Site #: 71025), Baltimore, Maryland
  - Boston Children's Hospital (Site #: 71001), Boston, Massachusetts
  - Helen DeVos Children's Hospital (Site #: 71035), Grand Rapids, Michigan
  - Washington University/St. Louis Children's Hospital (Site #: 71006), St Louis, Missouri
  - New York Medical College/Boston Children's Health Physicians, Westchester, New York
  - Duke University (Site #: 71033), Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center (Site #: 71017), Cincinnati, Ohio
  - Children's Hospital of Philadelphia (Site #: 71091), Philadelphia, Pennsylvania
  - UPMC Children's Hospital of Pittsburgh (Site #: 71008), Pittsburgh, Pennsylvania
  - Texas Children's Hospital (Baylor) (Site #: 71005), Houston, Texas
  - Seattle Children's Hospital (Site #: 71041), Seattle, Washington

REFERENCES:
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — http://www.niaid.nih.gov/about/dait